CLINICAL TRIAL: NCT04654104
Title: Predictive Role of Immune Checkpoints in COPD Evolution Towards Lung Cancer
Brief Title: Immune Checkpoints in COPD
Acronym: CP-COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Sanitaria Provinciale Di Catanzaro (Other); Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Principal Investigator, Clinical Professor, University of Catanzaro
Other Study IDs: 361/2020
Record Dates: First submitted 2020-11-20; First posted 2020-12-04 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Lung Cancer; Severe ARDS; Asthma; Copd
Keywords: systemic diseases
MeSH Terms: conditions — Lung Neoplasms; Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy never smokers: Clinical evaluation of immune check points expression. A prospective study
  Interventions: Other: check immune check points
- Smokers with normal lung function: evaluation of immune check points expression
  Interventions: Other: check immune check points
- Lung cancer: evaluation of immune check points expression
  Interventions: Other: check immune check points
- COPD: evaluation of immune check points expression
  Interventions: Other: check immune check points

INTERVENTIONS:
Other: check immune check points — we will evaluate the expression of immune check points

SUMMARY:
The aim of this study is to investigate the mechanisms underlying the complex interaction between Chronic obstructive pulmonary disease (COPD) and lung cancer. Therefore, in order to identify a possible role of immune checkpoints not only in the susceptibility to COPD development but also in its evolution towards lung cancer, will be evaluate the correlation between PD-L1 expression and cigarette smoke exposure in COPD patients.

Although there are many epidemiological studies highlighting the interconnections between COPD and lung cancer and the influence of cigarette smoke, the molecular bases of this association are less well defined. Initially they were thought to be driven just by innate inflammation, however, recent studies have also demonstrated the influence of the adaptive immune system. Despite this, the role of immune checkpoints in chronic lung inflammatory diseases such as COPD is less well understood. COPD is currently the 4th leading cause of death worldwide but is assessed to be the 3rd by the end of 2020 resulting in an economic and social burden that is in continuous progression.

DETAILED DESCRIPTION:
The aim of this study is to investigate the mechanisms underlying the complex interaction between Chronic obstructive pulmonary disease (COPD) and lung cancer. Therefore, in order to identify a possible role of immune checkpoints not only in the susceptibility to COPD development but also in its evolution towards lung cancer, will be evaluate the correlation between PD-L1 expression and cigarette smoke exposure in COPD patients.

Although there are many epidemiological studies highlighting the interconnections between COPD and lung cancer and the influence of cigarette smoke, the molecular bases of this association are less well defined. Initially they were thought to be driven just by innate inflammation, however, recent studies have also demonstrated the influence of the adaptive immune system. Despite this, the role of immune checkpoints in chronic lung inflammatory diseases such as COPD is less well understood. COPD is currently the 4th leading cause of death worldwide but is assessed to be the 3rd by the end of 2020 resulting in an economic and social burden that is in continuous progression.

Patients will be recruited from from the outpatient clinics of the Pulmonary and Critical Care Medicine department of "Mauro Scarlato" Hospital in Scafati, Italy in collaboration with the Operational Unit of Clinical Pharmacology and Pharmacovigilance of Catanzaro University.

171 patients will be divided according to the results of the anatomopathological examinations into four groups:

* Healthy never smokers
* Smokers with normal lung
* Cancer
* COPD (COPD group was divided in two subgroups: GOLD 1-2 group and GOLD 3-4 group).

ELIGIBILITY:
Inclusion Criteria:

* • over 18 years of age with suspected diagnosis of pulmonary neoplasia

  * signed the informed consent

Exclusion Criteria:

* • infected diseases

  * interstitiopathy
  * asthma,
  * autoimmune diseases,
  * neoplasia other than inclusion criteria
  * subjects on glucocorticoid therapy
  * alcohol consumption (>3 alcoholic beverages daily)
  * substance abuse
  * inability to give written informed consent
  * those who will not sign the consent to the processing of personal data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The levels of PD-1, PD-L1 and CTLA-4 will be evaluated by immunofluorescence and by RT-PCR on biopsy samples, which will be taken according to normal clinical practice. The checkpoint levels will be assessed before and after exposure after a medium of smoke also in the macrophages extracted from the BAL, which will be collected according to normal clinical practice, by RT-PCR.
  The aforementioned experiments will be carried out at the Pharmacology Section of the Department of Experimental Medicine, University of Campania Luigi Vanvitelli, their cost will not be borne by the NHS but will be fully borne by the aforementioned University.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
PD-L1 in bronchoalveolar lavage fluid | 1 month
  to evaluate the expression of PD-L1
CTLA-4 in bronchoalveolar lavage fluid | 1 month
  to evaluate the expression of CTLA-4
mucin-domain containing-3 (TIM-3) | 1 month
  to evaluate the expression of mucin-domain containing-3 (TIM-3) in bronchoalveolar lavage fluid
PD-1 in bronchoalveolar lavage fluid | 1 month
  to evaluate the expression of PD-1

SECONDARY OUTCOMES:
check point and smoke | 1 month
  to evaluate the correlation between PD-L1 expression and cigarette smoke exposure in COPD patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Luca Gallelli, Catanzaro, CZ
  - AO Materdomini, Catanzaro, Italia

IPD SHARING:
Plan to Share IPD: Yes
publication of the results
Supporting Information: Study Protocol, SAP
Time Frame: 12 months